CLINICAL TRIAL: NCT01543438
Title: Optimizing Emergency Aftercare With Mobile Video Prescriptions
Brief Title: Using Point-of-Care Video Prescriptions to Improve Aftercare Following Discharge From a Pediatric Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: healthEworks LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David J Mathison, Assistant Professor of Pediatrics & Emergency Medicine, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R41MD006695-01 (NIH)
Record Dates: First submitted 2012-02-22; First posted 2012-03-05 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Compliance; Emergency Department Aftercare; Emergency Department Utilization
Keywords: ED utilization; video education; mobile health; streaming media; underserved populations
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): current standard of care
- Intervention Group (Experimental): receives video prescription
  Interventions: Other: Video Prescription (additional education)

INTERVENTIONS:
Other: Video Prescription (additional education) — receives video prescriptions
  Arms: Intervention Group

SUMMARY:
The goal of this project is to develop the content and delivery platform that electronically distributes mobile video discharge education for underserved populations and to demonstrate utilization, satisfaction, and improved health outcomes.

DETAILED DESCRIPTION:
Emergency department (ED) visits have increased by 25% over the past decade. 85% of these patients are discharged, and the standard of care is to provide each patient/caregiver with written instructions that highlight how to care for a particular illness at home and signs to return to the hospital. Compliance with such ED discharge instructions is limited, leading to suboptimal medical care and unnecessary return visits to the ED. Inadequate health literacy, language disparities, and poor comprehension of written discharge information contribute to this problem. This health gap is more prevalent in children of young parents, low-income families, and minority populations where a disproportionate number of patients visit the ED for non-emergent care, often because of a lack of health education. The ED environment is chaotic and distracting and suboptimal to educate patients. Such education is best accomplished where aftercare occurs-in the home, but many patients lack direction and motivation to seek reliable sources of focused health education.

healthEworks LLC has developed Video Prescriptions™ - concise 3-5 minute video modules specific to the most common discharge diagnoses that patients receive in the ED. Further work is needed to develop a professional, diagnosis-specific product. These videos will feature Dr. Christina Johns, an emergency physician who specializes in delivering health information on camera. Each video will be interactive, high definition, designed for small screen size, such as for a smartphone or laptop computer. Each video prescription™ will highlight the transition from hospital to home and focuses on what the diagnosis means, how to treat it at home, and which signs should prompt the patient to return to the ED or seek urgent care. A HIPAA-compliant tablet-based platform will link ED patients with their personalized video education, establishing an innovative system of post-discharge information sharing.

The use of video prescriptions™ will improve patient health education for the 100 million patients who are discharged from U.S. ED's annually. This technology is particularly applicable for hospitals that face increasing pressures to provide performance measures for hospital discharge.

Video prescriptions™ will be utilized by ED patients, regardless of socioeconomic status, will improve patient satisfaction and reduce unnecessary ED return visits.

* Specific Aim 1: Demonstrate patient utilization of video prescriptions Criteria for acceptance: a hyperlink click rate of greater than 70%
* Specific Aim 2: Demonstrate improved health outcomes. Criteria for acceptance: a reduction in return visits by 10%
* Specific Aim 3: Demonstrate quality of video content by showing improved patient satisfaction scores. Criteria for acceptance: improvement in patient satisfaction scores by 20%

ELIGIBILITY:
Inclusion Criteria:

* fits one of diagnostic criteria
* not previously enrolled in past week

Exclusion Criteria:

* primary language other than english or spanish
* does not consent to receive email communication

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5000 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Video Prescription Utilization Rate | 6 months
  measured with hyperlink click rate and successful streaming verification

SECONDARY OUTCOMES:
ED Return Visit Rate | 6 months
  ED return visits within 72 hrs and one week. Will also be stratified into 'unnecessary' return visits by assessing resource use and billing data.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Medical Center (UMC and SZ campuses), Washington D.C., District of Columbia, United States